CLINICAL TRIAL: NCT04002089
Title: A Phase 1, Pilot, Open Label, Dose Escalation Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety, of EXPAREL Administered as Sciatic Nerve Block (In Popliteal Fossa), for Postsurgical Analgesia in Subjects Undergoing Bunionectomy
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety, of EXPAREL Administered as Sciatic Nerve Block (In Popliteal Fossa), for Postsurgical Analgesia in Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-122
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Bunion
MeSH Terms: conditions — Bunion | interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - EXPAREL (Experimental): A total of 10 subjects will be enrolled. Subjects in this cohort will receive 266mg of EXPAREL admixed with bupivacaine.
  Interventions: Drug: Exparel Injectable Product; Drug: Bupivacaine
- Cohort 2 - EXPAREL (Experimental): A total of 10 subjects will be enrolled. Subjects in this cohort will receive 133mg of EXPAREL admixed with bupivacaine.
  Interventions: Drug: Exparel Injectable Product; Drug: Bupivacaine
- Cohort 3 - EXPAREL (Experimental): A total of 10 subjects will be enrolled. Subjects in this cohort will receive 266mg of EXPAREL only
  Interventions: Drug: Exparel Injectable Product
- Cohort 4 - bupivacaine (Active Comparator): A total of 10 subjects will be enrolled. Subjects in this cohort will receive 100mg Bupivacaine only.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel Injectable Product — bupivacaine liposome injectable suspension
  Arms: Cohort 1 - EXPAREL; Cohort 2 - EXPAREL; Cohort 3 - EXPAREL
Drug: Bupivacaine — 1.3%, 13.3 mg/mL
  Arms: Cohort 1 - EXPAREL; Cohort 2 - EXPAREL; Cohort 4 - bupivacaine

SUMMARY:
This is a pilot, open label, single center study in 40 subjects undergoing bunionectomy. The study will assess and collect information on pharmacokinetics, pharmacodynamics, safety and efficacy of EXPAREL administered as a sciatic nerve block (in popliteal fossa).

A total of 10 subjects will be enrolled in each of the 4 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages 18 or older
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.
4. Body Mass Index ≥18 and ≤40 kg/m2

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (eg, amide-type local anesthetics, opioids, bupivacaine, NSAIDs)
2. Documented history of long-term diabetes or severe peripheral vascular disease
3. Renal (serum creatinine level >2mg/dL [176.8 μmol/L]) or hepatic dysfunction (serum alanine or aspartame transferase > 3 times the upper limit of normal).
4. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which, in the investigator's opinion may confound the post dosing assessments
5. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
6. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
7. Previous participation in an EXPAREL study
8. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance
9. Currently pregnant, nursing, or planning to become pregnant during the study
10. Clinically significant medical disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other conditions that would constitute a contraindication to participation in the study
11. Currently on neuroleptic agent [e.g., gabapentin, pregabalin (Lyrica), duloxetine (Cymbalta) etc.]
12. Inadequate sensory function on the foot (monofilament test)
13. Chronic opioid use in the last 30 days (≥30 morphine equivalents/ day)

    In addition, the subject may be withdrawn from the study if the subject meets the following criterion during or post-surgery:
14. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that, in the opinion of the investigator, renders the subject medically unstable or complicates the subject's post-operative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic 1 (Area under the plasma concentration) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1), 60(±2), 72(±2), 84(±2), 96(±3), 120(±3), 144(±3), and 168(±3) hours following block
  Area under the plasma concentration-versus-time curve (AUC).
Pharmacokinetic 2 (Cmax) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1h), 60(±2h), 72(±2h), 84(±2h), 96(±3h), 120(±3h), 144(±3h), and 168(±3h) hours following block
  Maximum plasma concentration (Cmax)
Pharmacokinetic 3 (half-life ) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1h), 60(±2h), 72(±2h), 84(±2h), 96(±3h), 120(±3h), 144(±3h), and 168(±3h) hours following block
  The apparent terminal elimination half-life (t1/2el).
Pharmacokinetic 4 (Apparent clearance) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1h), 60(±2h), 72(±2h), 84(±2h), 96(±3h), 120(±3h), 144(±3h), and 168(±3h) hours following block
  Apparent clearance (CL/F).
Pharmacokinetic 5 (volume of distribution) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1h), 60(±2h), 72(±2h), 84(±2h), 96(±3h), 120(±3h), 144(±3h), and 168(±3h) hours following block
  Apparent volume of distribution (Vd).
Pharmacokinetic 6 (Tmax) | predose (up to 15 min before block), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1h), 60(±2h), 72(±2h), 84(±2h), 96(±3h), 120(±3h), 144(±3h), and 168(±3h) hours following block
  Time of Cmax (Tmax)
Pharmacodynamic 1 (duration of sensory and motor block) | up to 15 min before block, 15 min(±5 min), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1), 60(±2), 72(±2), 84(±2), 96(±3), 120(±3), 144(±3), and 168(±3) hours following block
  Average duration of sensory block and motor block
Pharmacodynamic 2 (duration of sensory and motor block) | up to 15 min before block, 15 min(±5min), 30 min(±5min), 45 min(±5min), and 60 min (±15min) and 30 min(±5min), 45 min(±5min), 1(±15min), 2(±30min), 12(±30min), 24(±1), 60(±2), 72(±2), 84(±2), 96(±3), 120(±3), 144(±3), and 168(±3) hours following block
  Average duration of sensory block and motor block

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Nagaraj, Study Director — Medical Director
Locations (1):
- First Surgical Hospital, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: No